CLINICAL TRIAL: NCT03553004
Title: Niraparib in Metastatic Pancreatic Cancer After Previous Chemotherapy (NIRA-PANC): a Phase 2 Trial
Acronym: NIRA-PANC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-NIRA-PANC
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic pancreatic cancer; germline mutation; somatic mutation; Niraparib; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib Treatment (Experimental): * Niraparib 300 milligrams (mg) by mouth daily for 28 days (1 cycle = 28 days)
  * (Dose reduced to 200mg dose for participants whose baseline weight is less than 77 kilograms (kg) [169.756 pounds (lbs)] or baseline platelet count is less than 150,000 microliters (µL)).
  Interventions: Drug: Niraparib Treatment

INTERVENTIONS:
Drug: Niraparib Treatment — Niraparib treatment by mouth (oral)

SUMMARY:
The goal of this clinical research study is to learn if Niraparib can help to control metastatic pancreatic cancer. The safety of this drug will also be studied. Niraparib is FDA approved and commercially available for the treatment of ovarian cancer. Its use in this study is investigational.

ELIGIBILITY:
Key Inclusion Criteria:

* Screening tumor tissue analysis positive with germline or somatic mutation in genes involved in DNA repair.
* Ability of participant or Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent.
* Able to swallow oral study drug
* Histologically or cytologically confirmed adenocarcinoma of the exocrine pancreas
* Measurable disease
* Patients with history of other, non-pancreatic cancers with no evidence of active disease are eligible.
* Participants who have had any prior chemotherapy as first line and/or second line therapy for metastatic disease are eligible to seek enrollment. Patients who refuse chemotherapy or do not tolerate chemotherapy are eligible.
* Patients must have adequate organ function
* Women must have a negative serum pregnancy test within 72 hours to taking study treatment.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use approved forms of contraception prior to study entry, for the duration of study participation, and for 180 days following completion of therapy.

Key Exclusion Criteria:

* Patients simultaneously enrolled in any therapeutic clinical trial
* Patients have had investigational therapy administered within the past 4 weeks
* Current or anticipated use of other investigational agents while participating in this study.
* Patient has had prior treatment with a known poly polymerase inhibitor
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant, breast feeding or expecting to conceive children while receiving study treatment and for 180 days after the last dose of study treatment. There is a potential for congenital abnormalities and for this regimen to harm breast feeding infants.
* Patients must not have a known hypersensitivity to the components of niraparib or the excipients
* Patients must not have had major surgery within the last 3 weeks of starting the study and patient must have recovered from any effects of any major surgery
* Patients must not have had radiotherapy encompassing more than 20% of the bone marrow within 2 weeks or any radiation therapy within 1 week prior to Day 1 of protocol therapy
* Patients must not be immuno-compromised. Patients with splenectomy are allowed.
* Patients must not have received a transfusion (platelets or red blood cells) within 4 weeks of the first dose of study treatment
* Patients must not have current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study or interfere with the patient's participation for the full duration of the study treatment or that makes it not in the best interest of the patient to participate
* Patients must not have known, symptomatic brain or leptomeningeal metastases
* Patient must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 8 weeks
  Defined as the percentage of participants with overall response to therapy at 8 weeks, defined as Partial Response or Complete Response (PR + CR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 5 years
  Calculated as the percentage of participants with PFS from the time of initial study treatment until the time of progression, defined per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall Survival (OS) | Up to 5 years
  Calculated as the average length of time of survival from the time of initial study treatment until the time of death from any cause.
Disease Control | 8 weeks
  Calculated as the percentage of participants that achieve any of the following at 8 weeks: complete response, partial response, or stable disease, as defined by RECIST v1.1
Duration of Response | Up to 5 years
  Calculated as the average length of time between response to treatment and disease progression, defined per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Proportion of participants with adverse events (AEs) | Up to 5 years
  Defined per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Anup Kasi, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (6):
- United States (6):
  - University of Kansas Cancer Center - Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center - West, Kansas City, Kansas
  - University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freed IM, Kasi A, Fateru O, Hu M, Gonzalez P, Weatherington N, Pathak H, Hyter S, Sun W, Al-Rajabi R, Baranda J, Hupert ML, Chalise P, Godwin AK, A Witek M, Soper SA. Circulating Tumor Cell Subpopulations Predict Treatment Outcome in Pancreatic Ductal Adenocarcinoma (PDAC) Patients. Cells. 2023 Sep 13;12(18):2266. doi: 10.3390/cells12182266. PMID 37759489